CLINICAL TRIAL: NCT06935617
Title: Hiatus Hernia and Frailty
Brief Title: Hiatus Hernia in Old
Status: Completed | Type: Observational
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Tamer.A.A.M.Habeeb, prof of general surgery, laparoscopic and GIT surgery, Zagazig University
Other Study IDs: Hiatus hernia
Record Dates: First submitted 2025-04-13; First posted 2025-04-20 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Hiatus Hernia
MeSH Terms: conditions — Hernia, Hiatal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- hiatus hernia: HH operated by LNF
  Interventions: Procedure: nissein

INTERVENTIONS:
Procedure: nissein — nissein surgery

SUMMARY:
hiatus hernia in frail patient is common and requires suregry

DETAILED DESCRIPTION:
severe frail patients had high incidence of recurrence

ELIGIBILITY:
Inclusion Criteria:

* EP aged ≥60 years for giant sliding HH with

Exclusion Criteria:

* • who required a concurrent abdominal procedure at the same time as fundoplication (e.g., cholecystectomy)(n=5)

  * esophageal dysmotility(n=2)
  * progressive systemic sclerosis (n=1)

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: elderly pt with hh
Sampling Method: Non-Probability Sample
Enrollment: 266 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
recurrence | three years

IPD SHARING:
Plan to Share IPD: No